CLINICAL TRIAL: NCT02852590
Title: Relationship Between Adverse Drug Reactions and Unlicensed/ Off-label Drug Use in Hospitalized Children: an Observational Multicenter Prospective Study
Brief Title: Relationship Between Adverse Drug Reactions and Unlicensed/ Off-label Drug Use in Hospitalized Children
Acronym: EREMI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D21530
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Hospitalized Children
Keywords: Observational; Pediatric; Off-Label Use; Unlicensed drug use; Adverse Drug Reaction; Hospitalized Children; Pediatric inpatients
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Medications are the most commonly used clinical intervention and complications associated with their use are one of the most common causes of adverse events in health care. Adverse Drug Reactions (ADR) are a major cause of morbidity and pose a substantial burden on limited health care resources.

Many drugs used to treat children in hospitals are either not licensed for use in children or are prescribed outside the terms of their product license (off-label prescribing). This is mainly due to the lack of clinical trials in this vulnerable population, and both practical difficulties and ethical considerations arising from involving children in clinical research.

Drugs used within the specifications of the product license might be less likely to cause ADR compared to drugs that are either unlicensed or off-label for use in children. Few studies have shown a significant association between pediatric off-label drug use and ADR.

To compare the probability of ADR after a licensed drug prescription versus the probability of ADR after prescribing a drug off-label in children, we are conducting a multi-center prospective observational study in different pediatric hospital wards in France.

The availability of electronic health records made this study feasible. An automatic data extraction from hospital information systems has been implemented. A computer algorithm for determining pediatric drug labelling (i.e. off-label or unlicensed use) using the French summaries of product characteristics available in Thériaque® database has been developed. Detection of ADRs is carried out by health care professionals and research groups using a trigger tool and patients' electronic health records. The causality between ADRs and suspected medications is evaluated using the Naranjo and the French methods by regional pharmacovigilance centers. An independent pharmacovigilance board validates ADR evaluations, assesses both of their severity and avoidability, and indicates therapeutic alternatives to suspected medications.

This is, to our knowledge, the first large multi-center and prospective study in France that evaluates the relationship between adverse drug reactions and unlicensed/ off-label drugs use in hospitalized children. The results of this study will provide more information on the prescription practice and the amplitude, nature and consequences of unlicensed/off-label drug use in hospitalized children. It will also help identify the risk factors of ADR that could be used to implement preventive actions, and guide future research in the field. An indirect benefit is represented by the increase of physicians' awareness in detecting and declaring ADRs and by communicating the results to the health professionals and to the public. This study is funded by ANSM (the French Medicine Agency).

ELIGIBILITY:
Inclusion Criteria:

* Children from 0 to 15 years old [0 ; 15[ (including term and preterm newborn infants).
* Hospitalised for at least 3 days.
* Receiving at least one medication.

Exclusion Criteria:

* Children aged 15 to 18 years old [15 ; 18]
* Children hospitalized for an Adverse Drug Reaction or undergoing voluntary drug detoxification.
* Children who did not take any drugs during their hospital stay.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All eligible children will be recruited consecutively according to their hospital admission in the following wards : nephrology; hepato-gastroenterology; intensive care unit; endocrinology; child psychiatry; neurology; pneumology; pediatric cardiology; epilepsy, sleep and pediatric neurophysiology; general pediatrics.
Sampling Method: Non-Probability Sample
Enrollment: 6227 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
occurrence of an adverse drug reaction (ADR) | up to one month
  To compare the probability of occurrence of an adverse drug reaction (ADR) after a licensed prescription drug versus the probability of occurrence of an ADR after prescribing a drug off-label or unlicensed in patients aged 0-15 years hospitalized at least 3 days.

SECONDARY OUTCOMES:
proportion of pediatrics inpatients presenting at least one ADR | up to one month
  Compare the proportion of pediatrics inpatients presenting at least one ADR among inpatients with at least one off-labels or unlicensed prescription drug with the proportion of inpatients presenting at least one ADR among inpatients with all licensed prescription drugs
indications for which drugs are prescribed in term of licensed/ unlicensed/ off-label manner by age group | up to one month
Identify the factors influencing the risk of developing ADRs after prescribing a drug | up to one month
  These factors may include (but are not limited to) : age, gender, severity of the disease, concomitant treatments, number of administered medications, parenteral nutrition, prematurity, etc.
causality of ADRs | up to one month
  Physician Assessment
severity of ADRs | up to one month
  Physician Assessment
avoidability of ADRs | up to one month
  Physician Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Behrouz KASSAI, Pr, Principal Investigator — Pediatric Clinical Research and Investigation Centre CIC 1407 Inserm-UMR 5558 CNRS Lyon University & Hospices Civils de Lyon
Locations (1):
- Pediatric Clinical Research and Investigation Centre CIC 1407 Inserm-UMR 5558 CNRS Lyon University & Hospices Civils de Lyon, Lyon, France